CLINICAL TRIAL: NCT00722592
Title: A Randomized Phase II Trial Comparing EC145 and Pegylated Liposomal Doxorubicin (PLD/Doxil/Caelyx) in Combination, Versus PLD Alone, in Subjects With Platinum-Resistant Ovarian Cancer
Brief Title: Platinum Resistant Ovarian Cancer Evaluation of Doxil and Vintafolide (MK-8109, EC145) Combination Therapy (8109-009, EC-FV-04)
Acronym: PRECEDENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8109-009; EC-FV-04
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Ovarian Cancer
Keywords: cancer; ovarian; platinum-resistant; Phase II; EC145; EC20
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — EC145; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vintafolide + PLD (Experimental): Participants receive vintafolide 2.5 mg intravenous (IV) bolus on Days 1, 3, 5, 15, 17, and 19 and Pegylated Liposomal Doxorubicin (PLD) weight-based dose, IV on Day 1 of each 4-week cycle.
  Interventions: Drug: Vintafolide; Drug: pegylated liposomal doxorubicin (PLD); Other: EC20
- PLD Alone (Active Comparator): Participants receive PLD on Day 1 of each 4-week cycle.
  Interventions: Drug: pegylated liposomal doxorubicin (PLD); Other: EC20

INTERVENTIONS:
Drug: Vintafolide — 2.5 mg IV bolus on Days 1,3,5 and 15,17,19 of a 4-week cycle
  Other Names: EC145
  Arms: Vintafolide + PLD
Drug: pegylated liposomal doxorubicin (PLD) — 50 mg/m^2 (with dose based on ideal body weight for participants whose measured body weight is greater than their ideal body weight) intravenous infusion on Day 1 of a 4 week cycle. Dose reductions permitted for toxicity.
  Other Names: Doxil®; Caelyx®
Other: EC20 — During the screening period, participants at centers with EC20 imaging capability will receive a single intravenous injection of 0.1 mg EC20 labeled with 20-25 mCi technetium-99m followed by an imaging procedure. A second injection and imaging may be done after all therapy with the study drugs is done.
  Other Names: 99mTc-EC20

SUMMARY:
The objective of this study is to compare progression-free survival (PFS), based upon investigator assessment using Response Evaluation Criteria In Solid Tumors version 1.0 (RECIST 1.0) and clinical findings, in participants with platinum-resistant ovarian cancer who receive combination therapy with vintafolide and pegylated liposomal doxorubicin (PLD/Doxil®/Caelyx®) with that in subjects with platinum-resistant ovarian cancer who receive PLD alone.

DETAILED DESCRIPTION:
This is a Phase II clinical trial to evaluate the efficacy and safety of the combination of vintafolide and pegylated liposomal doxorubicin (PLD; available in the United States as Doxil® and outside the United States as Caelyx®) compared to PLD alone.

Vintafolide is a drug that is specifically designed to enter cancer cells via the folate vitamin receptor (FR). Experimental evidence shows that this target receptor is expressed on virtually all ovarian cancers. Early clinical evidence in a small number of Phase I subjects and in a subset of subjects in an on-going single-arm Phase II study suggests that vintafolide may have antitumor effect in women with advanced ovarian cancer and that it is generally well-tolerated. This evidence suggests that vintafolide may be useful as chemotherapy against advanced ovarian cancer.

Patients at centers with EC20 imaging capability will also undergo imaging with the folate receptor (FR-)targeting investigational diagnostic agent EC20 during the screening period to assess uptake of this agent into tumors. This non-invasive procedure will provide additional information on the utility of EC20 imaging to identify subjects with the FR molecular "target" before treatment with vintafolide therapy.

ELIGIBILITY:
Inclusion Criteria:

To qualify for randomization and treatment the following criteria must be met:

* Subjects must sign an approved informed consent form
* Subjects must be ≥ 18 years of age
* Subjects must have pathology-confirmed epithelial ovarian, fallopian tube, or primary peritoneal carcinoma
* Subjects must have platinum-resistant ovarian cancer, where platinum-resistant is defined as disease that responded to primary platinum therapy and then progressed within 6 months or disease that progressed during or within 6 months of completing secondary platinum therapy
* Subjects must have at least a single (RECIST-defined) measurable lesion on a radiological evaluation that is conducted no more than four weeks prior to beginning study therapy (EC145 and/or PLD).
* Subjects must have had prior debulking surgery
* Subjects must have received prior platinum-based chemotherapy but must not have received more than 2 prior systemic cytotoxic regimens. Subjects are allowed to receive, but are not required to receive, one additional non-cytotoxic regimen for the management of recurrent or persistent disease. Non-cytotoxic (biologic or cytostatic) agents include, but are not limited to, monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Subjects must have recovered (to baseline/stabilization) from prior cytotoxic therapy-associated acute toxicities. Subjects who have recovered from non-cytotoxic therapy-associated toxicity or who have "controlled" non-cytotoxic therapy toxicity (e.g., vascular endothelial growth factor-related hypertension) can be entered into the trial after a drug wash-out period of 4 half lives
* Subjects must have adequate organ function including:

  1. Bone Marrow Reserve: Absolute neutrophil count(ANC)≥ 1.5x10^9/L prior to treatment. Subjects on maintenance doses of granulocyte colony stimulating factor (G-CSF) are eligible. Platelets ≥ 100x10^9/L and hemoglobin ≥ 9 g/dL.
  2. Hepatic: Total bilirubin level < 1.5 x ULN and alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase(GGT), and alkaline phosphatase levels < 2.5 x ULN.
  3. Renal: Serum creatinine level ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min/1.73m^2 for subjects with serum creatinine levels above 1.5 x ULN.
  4. Cardiac: Left ventricular ejection fraction (LVEF) equal to or greater than

the institutional lower limit of normal. LVEF must be elevated within 90 days prior to Cycle 1 Day 1

* Subjects of childbearing potential must:

  1. Have a negative serum pregnancy test prior to initiation of the therapeutic regimen
  2. Practice an effective method of birth control (e.g., oral, transdermal or injectable contraceptives, intrauterine device, double-barrier contraception, such as diaphragm and spermicidal jelly) for the duration of their participation in the trial through 3 months following the last dose of study drug.

Exclusion Criteria:

The presence of any of the following will exclude the subject from the study:

* Diagnosis of tumor of low-malignant potential
* Prior exposure to PLD or anthracycline therapy
* Prior exposure to FR-targeted therapy (EC145, EC0225, farletuzumab, etc)
* Prior therapy with mouse antibodies
* Prior therapy with vinorelbine (Navelbine®) or vinca-containing compounds
* Prior abdominal or pelvic radiation therapy, radiation therapy to > 10% of the bone marrow, or prior radiation therapy within the past 3 years to the breast/sternum, dermal lesions, head or neck
* Recent (i.e., ≤ 6 weeks) history of abdominal surgery or peritonitis
* Serious comorbidities (as determined by the investigator) such as, but not limited to, active congestive heart failure or recent myocardial infarction. Subjects who require antifolate therapy for the management of comorbid conditions (e.g., rheumatoid arthritis) will be excluded from the trial.
* Pregnancy
* Concurrent malignancy or history of other cancer (except noninvasive skin cancer) within the last 5 years
* Symptomatic central nervous system metastasis
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy that is considered to be investigational (i.e., used for non-approved indications(s) and in the context of a research investigation). Use of low dose corticosteroid therapy (for nausea prophylaxis, etc) is acceptable; however, concomitant tamoxifen therapy is not. Supportive care measures are allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival based on investigator assessment using RECIST and clinical findings | Assessed within 12 months following completion of accrual

SECONDARY OUTCOMES:
Compare overall survival of subjects between the two treatment arms | Assessed within 18 months after initiation of PFS analysis
Evaluate the safety and tolerability of EC145 in combination with PLD | event driven
Compare objective response rate (ORR) and duration of response of EC145 in combination with PLD, versus PLD alone, based on investigator assessment when analyzed using RECIST. | event-driven
Explore the correlation between therapeutic response (e.g. PFS, radiologic response, etc) and 99mTc-EC20 levels | Assessed within 12 months following completion of accrual

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Naumann RW, Coleman RL, Burger RA, Sausville EA, Kutarska E, Ghamande SA, Gabrail NY, Depasquale SE, Nowara E, Gilbert L, Gersh RH, Teneriello MG, Harb WA, Konstantinopoulos PA, Penson RT, Symanowski JT, Lovejoy CD, Leamon CP, Morgenstern DE, Messmann RA. PRECEDENT: a randomized phase II trial comparing vintafolide (EC145) and pegylated liposomal doxorubicin (PLD) in combination versus PLD alone in patients with platinum-resistant ovarian cancer. J Clin Oncol. 2013 Dec 10;31(35):4400-6. doi: 10.1200/JCO.2013.49.7685. Epub 2013 Oct 14. PMID 24127448
- See also: Endocyte web site — http://www.endocyte.com